CLINICAL TRIAL: NCT06670703
Title: A Clinical Study of the Effects of Environmental Pollution on Obesity
Status: Active, not recruiting | Type: Observational
Sponsor: Dong Peng (Other)
Collaborators: Affiliated Hospital of Yunnan University (Other); The Second People's Hospital of Qujing (Unknown)
Responsible Party: Sponsor-Investigator, Dong Peng, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: ZZ2024-350-02
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Obesity and Overweight
Keywords: air pollution; obesity; prevalence; overweight; environment
MeSH Terms: conditions — Obesity; Overweight | interventions — Adiposity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- the obesity group: Obese patients attending the First Affiliated Hospital of Chongqing Medical University, the Affiliated Hospital of Yunnan University, and the Second People's Hospital of Qujing City.
  Interventions: Diagnostic Test: Obesity

INTERVENTIONS:
Diagnostic Test: Obesity — diagnosis as obese patients

SUMMARY:
This study aims to assess the effects of environmental pollution (including environmental indicators such as PM2.5, PM5, PM10, SO2, NOX, O3, and greening index) on obese patients and to explore the possible mechanisms by which environmental pollution promotes obesity.

DETAILED DESCRIPTION:
Firstly, the effects of environmental pollution on obese patients were investigated by analysing the baseline conditions and obesity levels (including BMI, waist circumference, hip circumference, etc.) and underlying diseases of obese patients in regions with different pollution levels. Secondly, the association between environmental pollution levels on blood test characteristics (including renal function, sex hormones, glucose tolerance test, trace elements, liver function and blood routine) of obese patients was investigated to find possible mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* obese patients with BMI ≥30;
* patients without surgical treatment prior to enrolment;
* willingness to participate in the study and sign an informed consent form;
* complete clinical data.

Exclusion Criteria:

* patients with systemic diseases such as severe cardiorespiratory insufficiency affecting the choice of treatment regimen;
* patients assessed by the investigator to be inappropriate for enrolment;
* patients with incomplete clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective observational study, which is expected to include patients diagnosed with obesity ( body mass index (BMI) ≥ 28 kg/m2).
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
incidence of obesity | From 18 years old until the developing obesity, through study completion, an average of 5 year.
  the time for overweight to obesity

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Affiliated Hospital of Yunnan University, Kunming, Yunnan
  - The Second People's Hospital of Qujing, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No
Ethics committees of the clinical centres where the studies were conducted did not allow the release of patient data.